CLINICAL TRIAL: NCT03734718
Title: The Role of Glucose-dependent Insulinotropic Polypeptide in the Pathological Glucose Homeostasis of Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: GIPHOT; H-18015379 (Other: Research Ethics in the Capital of Denmark)
Record Dates: First submitted 2018-10-22; First posted 2018-11-08 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Diabetes Mellitus, Type 1; Hypoglycemia
Keywords: Gastric Inhibitory Polypeptide; Diabetes Mellitus, Type 1; Hypoglycemia; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Glucagon; Incretin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases

STUDY DESIGN:
Intervention Model Description: placebo-controlled, double-blinded, cross-over study
Who Masked: Participant, Care Provider, Investigator
Masking Description: The peptides/placebo is prepared, in a randomized fashion, by a laboratory assistant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glucose-Dependent Insulinotropic Polypeptide (Active Comparator): 6-day continuous infusion of Glucose-Dependent Insulinotropic Polypeptide
  Interventions: Drug: GIP
- Placebo (Placebo Comparator): Saline
  Interventions: Drug: GIP

INTERVENTIONS:
Drug: GIP — Infusion of Glucose-dependent insulinotropic peptide

SUMMARY:
In the present project the investigators will evaluate whether glucagonotropic properties of the gut-derived incretin hormone glucose-dependent insulinotropic polypeptide (GIP) may be utilized as a safeguard against hypoglycemia in the daily life of participants with type 1 Diabetes

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 20 and 27 kg/m2
* T1D (diagnosed according to the criteria of the World Health Organization) with HbA1c <69 mmol/mol (<8.5%)
* Treatment with a stable insulin regimen ≥3 months
* T1D duration between 2 and 15years
* C-peptide negative (C-peptide ≤ 16 ng/ml)
* Informed consent

Exclusion Criteria:

* Anemia (hemoglobin outside normal range)
* Known liver disease and/or ALAT and/or ASAT > 2 times normal values
* Estimated glomerular filtration rate (eGFR) ≤60 ml/min/1.73 m2 or albuminuria
* Prior Cardiovascular events and/or abnormal heart rate/blood pressure
* Use of anti-diabetic medicine (other than insulin), corticosteroids or other drugs affecting glucose metabolism during the study period or within 30 days prior to randomization
* Any physical or psychological condition that the investigator feels would interfere with trial participation

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Caucasian men
Enrollment: 20 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Blood glucose | an average of 6 days
  Time spent in hypoglycemia, near-normoglycemia and hyperglycemia

SECONDARY OUTCOMES:
Incretin hormones | Evaluated at experimental day 0,1 and 6 of each intervention
  Incretin hormones GLP-1 and GIP. Incremental and total area under the Concentration-Time Curve
Free fatty acids (FFA) | Evaluated at experimental day 0,1 and 6 of each intervention
  Incremental and total area under the Concentration-Time Curve
Fat mRNA | At day 6, and 10 of the study
  mRNA analysis of fat biopsies
Fat Protein content | Evaluated at experimental day 0,1 and 6 of each intervention
  Protein analysis of fat biopsies
Blood pressure | The first 24 hours of intervention and at experimental day 6
  Changes in blood pressure, mm Hg
Pulse | The first 24 hours of intervention and at experimental day 6
  Changes in pulse, beats per minute
Glucose regulatory hormones | Evaluated at experimental day 0,1 and 6 of each intervention
  Counter regulatory hormones: glucagon, noradrenalin, cortisol, somatotropin, and insulin/c-peptide. Incremental and total area under the Concentration-Time Curve
Number of symptomatic hypoglycemic events | An average of 1 week
  Self-reported events

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center CopenhagenSteno Diabetes Center Copenhagen, Clinical Metabolic Physiology, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gilliam-Vigh H, Suppli MP, Heimburger SMN, Lund AB, Knop FK, Ellegaard AM. Cholesin mRNA Expression in Human Intestinal, Liver, and Adipose Tissues. Nutrients. 2025 Feb 8;17(4):619. doi: 10.3390/nu17040619. PMID 40004948
- [Derived] Heimburger SMN, Hoe B, Nielsen CN, Bergman NC, Skov-Jeppesen K, Hartmann B, Holst JJ, Dela F, Overgaard J, Storling J, Vilsboll T, Dejgaard TF, Havelund JF, Gorshkov V, Kjeldsen F, Faergeman NJ, Madsen MR, Christensen MB, Knop FK. GIP Affects Hepatic Fat and Brown Adipose Tissue Thermogenesis but Not White Adipose Tissue Transcriptome in Type 1 Diabetes. J Clin Endocrinol Metab. 2022 Nov 25;107(12):3261-3274. doi: 10.1210/clinem/dgac542. PMID 36111559
- [Derived] Heimburger SMN, Hoe B, Nielsen CN, Bergmann NC, Hartmann B, Holst JJ, Vilsboll T, Dejgaard TF, Christensen MB, Knop FK. The effect of 6-day subcutaneous glucose-dependent insulinotropic polypeptide infusion on time in glycaemic range in patients with type 1 diabetes: a randomised, double-blind, placebo-controlled crossover trial. Diabetologia. 2021 Nov;64(11):2425-2431. doi: 10.1007/s00125-021-05547-8. Epub 2021 Aug 17. PMID 34405256